CLINICAL TRIAL: NCT02333344
Title: The Efficacy Study of Aclasta (Zoledronic Acid 5mg) on Prosthetic Fixation in Postmenopausal Women After Cementless Total Hip Arthroplasty (THA): a 24 Months, Single Center, Open- Label, Randomized, Parallel Controlled Study
Brief Title: The Efficacy Study of Aclasta on Prosthetic Fixation in Postmenopausal Women After THA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant, for strategic reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HCN13
Record Dates: First submitted 2014-10-12; First posted 2015-01-07 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Prosthetic Fixation After Cementless Total Hip Arthroplasty
Keywords: prosthetic fixation
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic acid 5mg (Experimental): interventional group which receive yearly Zoledronic acid 5mg/100ml infusion treatment for two years
  Interventions: Drug: Zoledronic acid 5mg
- blank (No Intervention): blank group

INTERVENTIONS:
Drug: Zoledronic acid 5mg — two-year Zoledronic acid 5mg infusion treatment
  Other Names: aclasta
  Arms: Zoledronic acid 5mg

SUMMARY:
It's to investigate the efficacy of Zoledronic acid treatment on the early prosthetic fixation in post-menopausal osteoporosis women under cementless total hip arthroplasty after 24-month observation.

DETAILED DESCRIPTION:
To investigate the efficacy of Zoledronic acid and placebo treatment on the prosthetic transverse translation in post-menopausal osteoporosis women under cementless total hip arthroplasty by Radiostereometry （RSA）in two-year follow-up period .

Meanwhile to assess efficacy of Zoledronic acid treatment on the vertical translation of acetabulum and the subsidence translation of femoral stem by Radiostereometry（RSA), prevention of peri- prosthetic bone loss by observing the local average bone mineral density ( BMD ) changes for 7 femoral region Gruen zones through Dual Energy X-ray Absorptiometry (DXA）scans, et al.

ELIGIBILITY:
Inclusion Criteria:

Patients who was diagnosed with Post-menopausal osteoporosis( bone mineral density T<-2.5;or with previous fragility fracture, bone mineral density T -2.5~-1.5), responding to Zoledronic acid, within one week after the successful cementless total hip arthroplasty surgery.

Exclusion Criteria:

1. Patients with any history of disorders except osteoporosis known to severely affect bone and mineral metabolism such as Paget disease;
2. Patients who suffer from secondary osteoporosis
3. Patients who were treated with bisphosphonate within the previous one year ,anabolic drug or strontium;
4. Patients with contraindications for Zoledronic acid:
5. Patients with invasive malignant tumor on any organ in the past 5 years, treated oruntreated;
6. Patients with primary hyperparathyroidism.
7. Serum calcium >2.75mmol/L (11.0mg/dL).
8. Patients who are unwilling to accept the treatment of Zoledronic acid.
9. Patients who accepted the treatment of investigational product and/or device in the 30 days before randomization.
10. Patients with any medical or mental diseases, which prevent patients from complying with protocols or completing protocols, judged by investigators.
11. Patients with the medical history of inflammation of the iris or uveitis, except the inflammation which is secondary to trauma and cured 2 years ago before screening.
12. Patients with the medical history of diabetic nephropathy or diabetic retinopathy.
13. Patients aged under 60 years old and whose result of urine pregnancy test paper is positive.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2020-01-28 (Estimated); Study Completion 2020-01-28 (Estimated)

PRIMARY OUTCOMES:
the transverse translation (μm) | baseline and month12,month 24
  the transverse translation (μm, outside-inside) between acetabular prosthesis markers and reference point

SECONDARY OUTCOMES:
average bone mineral density ( BMD ) | 1w,6m,12m and 24m after THA operation
  the local average bone mineral density ( BMD ) changes for 7 femoral region Gruen zones through Dual Energy X-ray Absorptiometry （DXA）scans.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Shanghai, Shanghai Municipality, China